CLINICAL TRIAL: NCT06525090
Title: Investigation of the Psychometric Properties of the Turkish Child-Friendly Oral Health Questionnaire
Brief Title: Turkish Version of Child-Friendly Oral Health Questionnaire
Status: Completed | Type: Observational
Sponsor: Muğla Sıtkı Koçman University (Other)
Collaborators: recep kara (Unknown); özgül Cartı Dörterler (Unknown); gülay manav (Unknown)
Responsible Party: Principal Investigator, Gonca Karayagiz Muslu, Associate Professor, Muğla Sıtkı Koçman University
Record Dates: First submitted 2024-07-23; First posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Tooth Diseases; Oral Disease
Keywords: validity; reliability; oral health
MeSH Terms: conditions — Tooth Diseases; Mouth Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 298 school children aged 9-10 years: 298 school children aged 9-10 years.
  Interventions: Other: no intervention-child-administered questionnaires

INTERVENTIONS:
Other: no intervention-child-administered questionnaires — The implementation of the research was started after getting approval from Mugla Sıtkı Kocman University Health Sciences Ethics Committee and TR Ministry of National Education Research, Competition and Social Activity. The purpose of the study was explained by the researchers to the administrators of the schools where the study was conducted and planning was made with the school administration. The data were collected in 15-20 minutes from the students who agreed to participate in the study during the course hours deemed appropriate by the administration. The purpose of the study and how to fill in the measurement tools was explained to the students, and it was stated that the research data would be kept confidential and used only by the researcher. The self-administered questionnaires were filled out on the paper. Verbal consent was obtained from the students participating in the study and written informed consent was obtained from their parents.

SUMMARY:
Oral problems are a common occurrence among school-age children. In order to develop effective oral health interventions and services, it is essential to determine children's oral health behaviours using an internationally accepted standardised instrument that is child-friendly. However, no instrument currently exists to measure oral health according to the Theory of Planned Behaviour (TPB) in Turkish school-aged children. The aim of this study was to investigate the psychometric properties of the Oral Health Questionnaire, which includes the components of the theory of planned behavior such as attitude toward children's oral health, subjective norm, perceived behavioral control, and self-efficacy, for the Turkish population

DETAILED DESCRIPTION:
The Oral Health Questionnaire was used as the data collection tool in the study. It was developed by Davison et al. (2017) as a child-friendly scale consisting of 57 questions in a 5-point Likert type based on the TPB [6]. The scale consists of three parts. The first part consists of questions to obtain sociodemographic information (items 1-9), and the second part consists of questions to determine the behavioral characteristics of the individual toward tooth brushing. Tooth brushing behaviors are evaluated based on the individual's statements. The last part of the scale consists of questions to determine direct and indirect measures of beliefs based on the theory of planned behavior. We used the Pictorial rating Likert scales as original.

The translation is the first step in the adaptation process. After the scale was translated into Turkish, a common Turkish version was developed by the researchers through group work. The Turkish version of the scale was translated into English by a different linguist who is an expert in both Turkish and English. To determine the content validity of the scale whose language validity was completed, it was submitted to the opinions of 10 faculty members, including pediatric nursing, public health nursing, and pedodontics experts. After receiving expert opinions, it is recommended to administer the scale to a group of approximately 20-30 individuals who have similar characteristics with the study subjects for pilot study. For the language validity of the scale, the translation-back translation technique was used, and for content validity, I-CVI and S-CVI were used Davis technique. According to Davis technique, each item of the scale was evaluated by ten faculty members who are experts in the field by choosing one of the four rating options from 1 (not relevant) to 4 (highly relevant). Item Content Validity Index (I-CVI) for each item was obtained by dividing the number of experts who chose option (3) or (4) when evaluating each item and dividing by the total number of experts. The intraclass correlation coefficient was used to evaluate the expert opinions for the content validity of the scale. Regarding reliability, the Cronbach alpha reliability coefficient was used to evaluate the internal consistency of the scale and its sub-dimensions, and Pearson product-moment correlation was used to compare item-total score correlations. Correlation and regression analysis were conducted for predictive validity. While the sample size was analyzed with Kaiser-Meyer-Olkin, its suitability for factor analysis was tested with Bartlett's Test of Sphericity, factor analysis, and principal component analysis. CFA was used to determine whether the items and subscales explained the original scale structure. CFA were performed on the same sample, the general sample was randomly split. The model verification of the comparative fit index (CFI) was conducted based on the chi-square test, degree of freedom, root mean square error of approximation (RMSEA), goodness of fit index (GFI), and normal fit index (NFI)

ELIGIBILITY:
Inclusion Criteria:

* Third-class students of central primary schools affiliated with the Directorate of National Education in Fethiye,
* Those without any communication barrier
* Those with reading and writing skills who can answer questionnaires
* Families who agreed to participate in the study and students who volunteered

Exclusion Criteria:

* Students and the parents who did not agree to participate in the study or who wanted to leave the study after it started were excluded from the study

Ages: 9 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The population of the study consisted of 5077 primary school students studying in 12 primary schools in the center of Fethiye in the 2020-2021 academic year. The study population comprised students in the third class of all primary schools in the centre of Fethiye. It is well-established that the sample size in validity and reliability studies should be at least 3-10 times the number of items.[11] To ensure the homogeneous distribution of students, the stratified random sampling method was used. In the sample determined by the stratified random sampling method, the number of students per school was determined and the students in the schools were stratified according to their classes, and data were collected from a total of 298 students
Sampling Method: Probability Sample
Enrollment: 298 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
reliability | 2 months
  To measure stability of the test over time by Turkish Version of Child-Friendly Oral Health Questionnaire. Turkish Version of Child-Friendly Oral Health Questionnaireis filled with two week interval.
validity | 6 months
  To test in order to establish the correlation among the proposed instrument and instruments that had already been translated and validated. factor analysis was done.

CONTACTS AND LOCATIONS:
Locations (1):
- 12 Primary Schools, Fethiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided